CLINICAL TRIAL: NCT06571123
Title: The Effect of Interactive Floor on Postoperative Pain and Mobilization of Children; Randomized Controlled Trial
Brief Title: The Effect of Interactive Floor on Postoperative Pain and Mobilization of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Huriye Karadede, Lecturer, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IstanbulAU Nursing Department
Record Dates: First submitted 2024-08-13; First posted 2024-08-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain Management
Keywords: Postoperative pain; pediatric surgery; nursing care; technology-based approach; mobilization; Interactive floor
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: group using interactive floor (Experimental): Postoperative mobilization of children in this group will be provided on the interactive floor installed in the relevant ward.
  Interventions: Other: İnteractive floor
- Control Group (No Intervention): The postoperative mobilization of children in this group will be provided in the corridor, which is the routine of the relevant service, and they will be prevented from seeing the interactive floor before mobilization. Children in this group will be allowed to use the interactive floor in their mobilization after their 3rd mobilization.

INTERVENTIONS:
Other: İnteractive floor — Interactive floor The interactive floor system includes a computer, camera and projection. With the projection, videos that are ready on the computer are projected on the floor, image processing is done with the camera and it detects whether there is an object on the floor or not and creates effects on the video. For example, on the floor containing colored balloons, the balloons burst with the movement of the child. With this visual mobility, it is aimed to draw the child's attention to another direction.
  Arms: Experimental Group: group using interactive floor

SUMMARY:
This research is planned to examine the effect of "interactive floor" on post-operative pain and mobilization in children within the scope of diversion method.

Research Question: Does the interactive floor affect children's post operative pain and mobilization?

Hypotheses of the Study:

H0: There is no difference between the postoperative pain score and mobilization time of children mobilized on the interactive floor and children mobilized with routine applications.

H1: Children mobilized on the interactive floor have lower pain scores than children in the control group.

H2: Children mobilized on the interactive floor have longer mobilization times than children in the control group.

H3: Children mobilized on the interactive floor have lower peak heart rate than children in the control group.

H4: Oxygen saturation of children mobilized on the interactive floor is higher than children in the control group.

DETAILED DESCRIPTION:
Pre-Mobilization:

The data for the child and family in the Interactive floor group and the control group who agreed to participate in the study and whose consent was obtained will be recorded by the researcher in the 'Child and Family Introductory Information Form' before mobilization with the patient file and face-to-face interview technique. Immediately before the 1st, 2nd and 3rd mobilizations of the child participating in the study in the postoperative period, pain score, peak heart rate and oxygen saturation values will be recorded without the child getting out of bed (while resting in bed).

During Mobilization:

Experimental group: Mobilization of children in this group will be provided on the interactive floor installed in the relevant ward. During the 1st, 2nd and 3rd mobilization, the child will be accompanied by the parent, nurse and researcher. In addition, during the 1st, 2nd and 3rd mobilization (the mobilization time will be evaluated by taking into account the time from the child getting out of bed to returning to bed), the mobilization time of the children will be measured with a stopwatch by an observer nurse who is not involved in the study and recorded in the data collection form. The mobilization time will depend on the child's own will and no restrictive intervention will be made by the researcher. In addition, pain scores, peak heart rate and oxygen saturation values will be recorded during the 1st, 2nd and 3rd mobilization (after the child has finished walking and before/while standing on the bed).

Control group: Mobilization of children in this group will be provided in the corridor, which is the routine of the relevant service, and they will be prevented from seeing the interactive floor before mobilization. Children in this group will be allowed to use the interactive floor in their mobilization after their 3rd mobilization.

During mobilization, the child will be accompanied by his/her parent, nurse and researcher. During the 1st, 2nd and 3rd mobilization, the child will be accompanied by his/her parent, nurse and researcher. In addition, during the 1st, 2nd and 3rd mobilization (the mobilization time will be evaluated by considering the time from the time the child gets out of bed to the time the child returns to bed), the mobilization time of the children will be measured with a stopwatch by an observer nurse who is not involved in the study and recorded in the data collection form. The mobilization time will depend on the child's own will and no restrictive intervention will be made by the researcher. In addition, pain score, peak heart rate and oxygen saturation values will be recorded during the 1st, 2nd and 3rd mobilization (after the child has finished walking and before/while standing on the bed).

After Mobilization: Immediately after the 1st, 2nd and 3rd mobilizations of the children in both groups, pain scores, peak heart rate and oxygen saturation values of the children will be recorded when the child sits/ lies down on the bed and after the children rest in the bed for 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Speak and understand Turkish
* Children whose parents agreed to participate in the study,
* Between 3 and 6 years old,
* Mobilization for the first time after surgical intervention
* No previous experience with other surgical procedures
* Ability to walk independently
* Children with vesico-uretero renal reflux, torsion of the ovarian pedicle of the ovary and fallopian tube, hypospadias, hirschsprung's disease, undescended testis, persistent cloaca, hydronephrosis, ureteropelvic junction obstruction, appendicitis, anus atresia/stenosis/fistula, biliary atresia, circumcision, phimosis and paraphimosis, post-traumatic surgery

Exclusion Criteria:

* Daily surgical procedures performed
* Having a health problem that prevents him/her from walking
* Serious complications after the operation
* Having any visual, auditory and mental problems
* The physician reports a problem that may prevent him/her from walking

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score | The child will be asked to rate the Wong-Baker FACES Pain Rating Scales 3 times: immediatelybefore mobilization, during mobilization and immediately after the mobilization.
  Wong-Baker FACES Pain Rating Scale The Wong-Baker Faces Pain Rating Scale is a pain scale that was developed by Donna Wong and Connie Baker. The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain.
  There are 6 faces in the Wong-Baker Pain Scale. The first face represents a pain score of 0, and indicates "no hurt". The second face represents a pain score of 2, and indicates "hurts a little bit". The third face represents a pain score of 4, and indicates "hurts a little more". The fourth face represents a pain score of 6, and indicates "hurts even more". The fifth face represents a pain score of 8, and indicates "hurts a whole lot"; the sixth face represents a pain score of 10, and indicates "hurts worst". This pain scale was originally developed for children.

SECONDARY OUTCOMES:
Mobilization Time | 1st, 2nd and 3rd postoperative mobilization of the child. Each mobilization will take an average of 5-15 minutes.
  Duration of the child's 1st, 2nd and 3rd postoperative mobilization The study is planned to be conducted at the first (approximately 8 hours after surgery), second (approximately 9 hours after surgery) and third (approximately 10 hours after surgery) postoperative mobilization of the children.

CONTACTS AND LOCATIONS:
Overall Officials: Huriye Karadede, Principal Investigator — Istanbul Aydın University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University Cerrahpaşa Cerrahpasa Faculty of Medicine, Bakırköy, Istanbul
  - Istanbul Aydin University, Istanbul, Istanbul

IPD SHARING:
Plan to Share IPD: No
I don't want to mislead you as I'm just starting my research.

REFERENCES:
- [Result] Topcu SY, Semerci R, Kostak MA, Guray O, Sert S, Yavuz G. The effect of an interactive robot on children's post-operative anxiety, mobilization, and parents' satisfaction; randomized controlled study. J Pediatr Nurs. 2023 Jan-Feb;68:e50-e57. doi: 10.1016/j.pedn.2022.11.009. Epub 2022 Nov 24. PMID 36437131